CLINICAL TRIAL: NCT07310186
Title: Salvage Treatment Strategies and Clinical Outcomes in Diffuse Large B-cell Lymphoma After Failure of Polatuzumab Vedotin-based Combination Therapy: A Multi-center, Retro- and Prospective, Observational, Real-World Study
Brief Title: Treatment and Outcomes of DLBCL After Progression on Polatuzumab Vedotin-based Combination Therapy
Status: Not yet recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PUMCH-NHL-022
Record Dates: First submitted 2025-07-22; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-07

CONDITIONS: Diffuse Large B Cell Lymphoma (DLBCL)
Keywords: DLBCL; polatuzumab vedotin; Salvage Treatment
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: observational study — this is an observational study, we do not interfere with treatment strategies

SUMMARY:
Diffuse Large B-cell Lymphoma (DLBCL) is a common hematologic malignancy. Even after standard first-line treatment, approximately 40% of patients will experience relapse. Currently, polatuzumab vedotin (pola) has been incorporated into DLBCL treatment (both for newly diagnosed and relapsed cases). However, for patients whose disease progresses after pola-containing regimens, the subsequent treatment options, efficacy, and survival outcomes remain unclear. Understanding these real-world scenarios is of great significance, as it can guide clinicians in developing better and more tailored treatment strategies for patients in the future.

Therefore, we plan to conduct this real-world study titled "Salvage Treatment Strategies and Clinical Outcomes in Diffuse Large B-cell Lymphoma After Failure of Polatuzumab Vedotin-based Combination Therapy", aiming to obtain real-world data from the Chinese population.

DETAILED DESCRIPTION:
This is a retro- and prospective, observational study

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with DLBCL
* Age ≥18 years
* Prior treatment with a polatuzumab vedotin (pola)-containing regimen and confirmed disease progression (refractory/relapsed) after this therapy.
* Availability of complete electronic medical records and ability to be contacted via telephone.
* Full understanding of the study, voluntary participation, and willingness to sign the informed consent form.

Exclusion Criteria:

* Patients who have not received pola-based regimen treatment.
* Incomplete electronic medical records or unreachable by telephone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 200
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
complete response rate | through study completion, an average of 2 years
  the ratio of patients achieves complete response